CLINICAL TRIAL: NCT00434135
Title: A Phase II Randomized Trial Assessing the Combination of Gemcitabine and Pemetrexed in the First Line Treatment of Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Alimta and Gemcitabine in Non-Small Cell Lung Cancer
Acronym: ANGEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Italy Cooperative Oncology Group (Other)
Responsible Party: Pasquale Comella MD, Southern Italy Cooperative Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SICOG trial 0506
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Non-Small Cell Lung Cancer; Stage IIIB or IV
Keywords: gemcitabine; pemetrexed; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gemcitabine 1,250 mg/sqm days 1 and 8 + Alimta 500 mg/sqm day 8, every 3 weeks
  Interventions: Drug: gemcitabine plus pemetrexed, paclitaxel plus gemcitabine
- B (Active Comparator): Paclitaxel 120 mg/sqm days 1 and 8 + Gemcitabine 1,000 mg/sqm days 1 and 8, every 3 weeks
  Interventions: Drug: gemcitabine plus pemetrexed, paclitaxel plus gemcitabine

INTERVENTIONS:
Drug: gemcitabine plus pemetrexed, paclitaxel plus gemcitabine — gemcitabine 1,250 mg/sqm days 1&8 + pemetrexed 500 mg/sqm day 8 paclitaxel 120 mg/sqm + gemcitabine 1,000 mg/sqm days 1&8

SUMMARY:
The aims of this study are: (1) to assess the safety and activity of gemcitabine plus Alimta (pemetrexed) regimen (GA regimen) in patients with advanced NSCLC patients in the context of a randomized trial, and (2) to compare the GA with the paclitaxel plus gemcitabine (PG regimen) in terms of toxicity and QoL

DETAILED DESCRIPTION:
Patients with stage IIIB or IV non-small cell lung cancer will be randomly allocated to receive: (a)PG regimen: paclitaxel 120 mg/sqm followed by gemcitabine 1,000 mg/sqm i.v. on days 1 & 8 q 3 weeks; (b)GA regimen: gemcitabine 1,250 mg/sqm i.v. on day 1 (plus folinic acid 350 μg daily orally and vitamin B12 1,000 μg i.m. q 9 weeks), pemetrexed (Alimta®) 500 mg/sqm i.v. on day 8 followed by gemcitabine 1,250 mg/sqm, q 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed locally advanced (stage IIIB) or metastatic (stage IV) NSCLC
2. No previous adjuvant or palliative chemotherapy
3. No previous radiotherapy
4. Presence of at least one unidimensionally measurable lesion (Appendix 2)
5. ECOG performance status of 0 or 1 (Appendix 3)
6. Charlson score ≤ 2 (Appendix 4)
7. Adequate bone marrow function (absolute neutrophil count ≥ 2 x 109/L, platelet count ≥ 100 x 109/L, and hemoglobin level ≥ 100 g/L), and adequate liver function (bilirubin level < two times the upper limit of normal, AST and/or ALT < three times the upper limit of normal, prothrombin time < 1.5 times control), and creatinine clearance ≥ 60 ml/min.
8. Absence of symptomatic CNS metastases (patients with cerebral metastases treated with brain irradiation may be included), severe cardiac arrhythmia or heart failure, second or third degree heart block or acute myocardial infarction within 4 months prior to study entry.
9. No major surgery or pleurodesis within 14 days prior to enrollment.
10. Life expectancy of at least 12 weeks.
11. No previous or concurrent malignancy, except inactive non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer if the patient has been disease-free for more than 5 years.
12. Written informed consent

Exclusion Criteria:

1. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease).
2. Patients with clinically significant effusions.
3. Any other malignancies within 5 years that could affect therapy evaluation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Response rate of patients treated with the gemcitabine plus Alimta regimen | after 3 cycles

SECONDARY OUTCOMES:
Safety of patients treated with gemcitabine plus Alimta regimen | at the end of treatment
Quality of life of patients treated with gemcitabine plus Alimta regimen | after 3 cyces

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Comella, MD, Principal Investigator — National Tumor Institute, Naples, Italy
Locations (1):
- National Tumor Institute, Naples, Italy